CLINICAL TRIAL: NCT01539707
Title: A Multicenter, Open-label, Single-dose Study to Evaluate Pharmacokinetics, Safety and Tolerability of Solifenacin Succinate Suspension in Pediatric Subjects From 5 to Less Than 18 Years of Age With Neurogenic Detrusor Overactivity (NDO)
Brief Title: Single Dose Study to Measure Blood Levels and Safety of a Drug for Children With Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 905-CL-079; 2011-000250-28 (EudraCT Number)
Record Dates: First submitted 2012-02-07; First posted 2012-02-27 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Overactive Bladder; Neurogenic Detrusor Overactivity
Keywords: Solifenacin succinate suspension; Pharmacokinetics; Phase 1; Neurogenic Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AD-PED 5 mg (Experimental): Male and female adolescents aged 12 to less than 18 years old who receive pediatric equivalent dose (PED) of 5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 5 mg
- CH-PED 5 mg (Experimental): Male and female children aged 5 to less than 12 years old who receive PED of 5 mg of solifenacin succinate.
  Interventions: Drug: Solifenacin succinate suspension 5 mg

INTERVENTIONS:
Drug: Solifenacin succinate suspension 5 mg — Adolescents and children are given a single dose of solifenacin succinate liquid suspension orally via syringe in the morning of day 1 followed by a glass of water. Doses are calculated per weight of the participant, targeting to have equivalent dose of 5 mg dose of solifenacin once daily in adults (referred to as PED of 5 mg).
  Other Names: YM905

SUMMARY:
The purpose of this study is to evaluate blood levels of solifenacin succinate (the study drug) in children with neurogenic detrusor overactivity after taking a single oral dose. If the bladder contracts strongly and without warning, the muscles surrounding the urethra (detrusor muscles) may not be able to keep urine from passing. This may happen as a consequence of spinal cord defects, and then is called neurogenic detrusor overactivity.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of NDO, confirmed by urodynamics
* Weight and height are within normal percentiles (3rd to 97th percentile) according to Centers for Disease Control and Prevention (CDC) growth charts
* Subject's bowel function is being actively managed
* Able to swallow the study medication in accordance to the protocol
* Female subjects of childbearing potential and sexually active agree to use a reliable form of birth control for the duration of the study and for at least one month after ending study treatment. Sexually active male subjects agree to use a barrier method of birth control for the duration of the study and for at least one month after ending study treatment
* Subject and subject's parent(s)/legal guardian are willing and able to comply with the study requirements and with the concomitant medication restrictions

Exclusion Criteria:

At screening:

* Subject is breastfeeding or pregnant. Subjects of childbearing potential must have a negative serum pregnancy test
* Subject with any of the following gastrointestinal (GI)conditions: partial or complete bowel obstruction, decreased motility (e.g., paralytic ileus) or at risk for gastric retention
* Current fecal impaction or history of hospitalization for fecal impaction with enema in the past 2 years
* History of QTc prolongation or risk of QT prolongation (e.g., hypokalemia, family history of Long QT Syndrome [LQTS]). QT interval greater than 470 ms at baseline
* Any clinically significant abnormality on ECG
* History or current diagnosis of any malignancy
* Diagnosis of central or X chromosome-linked diabetes insipidus
* Cystatine C is greater than or equal to 2 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is greater than or equal to 2 times the ULN or total bilirubin greater than or equal to 1.5 times the ULN
* Any other clinically significant out of range results of urinalysis, biochemistry or hematology
* Known or suspected hypersensitivity to solifenacin (or other anticholinergics), any of the excipients used in the current formulation or previous severe hypersensitivity to any drug
* Subject has participated in another clinical trial and/or has taken an investigational drug within 30 days (or 5 half-lives of the drug whichever is longer) prior to Day 1
* Requires ongoing treatment with any of the following prohibited medications: antimuscarinic therapy, tricyclic/tetracyclic antidepressants, H1 antihistamines, strong CYP3A4 inhibitors, strong CYP3A4 inducers (many antiepileptic drugs like carbamazepine, phenytoin and phenobarbital)
* Mean systolic blood pressure greater than the 95th percentile according to age and height and/or greater than 140 mmHg [National Institute of Health, 2005], judged as clinically significant by the investigator
* Subject's parent(s)/legal guardian is an employee of the Astellas Group, the Contract Research Organization (CRO) involved, or the investigator site executing the study

At Day 1:

* Consumption of grapefruit and products made of it (e.g., juice), and Seville oranges and products made of it (e.g., marmalade) within 14 days prior to Day 1
* Positive drug screen test for drugs of abuse at Day 1
* Positive alcohol breath test at Day 1
* Use of prohibited prior and concomitant medication:

  * Antimuscarinics, tricyclic/tetracyclic antidepressants, H1

antihistamines within 5 half-lives prior to intake of study drug at Day 1

* Prescribed or over the counter (OTC) drugs that are potent cytochrome P450 (CYP) 3A4 inhibitors (e.g., ketoconazole), CYP3A4 substrates with higher affinity (e.g., verapamil, diltiazem), or potent CYP3A4 inducers (e.g., rifampicin, phenytoin, carbamazepine), including natural and herbal remedies (e.g., St. John's Wort) within 14 days prior to intake of study drug at Day 1

  * Donation of blood or blood products within 3 months prior to Day 1.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2012-08-13 (Actual); Study Completion 2012-08-13 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | Day 1 predose up to Day 7 postdose
Time to Attain Cmax (tmax) | Day 1 predose up to Day 7 postdose
Area Under the Concentration-time Curve Extrapolated to Infinity (AUCinf) | Day 1 predose up to Day 7 postdose
Apparent Terminal Elimination Half-life (t1/2) | Day 1 predose up to Day 7 postdose
Apparent Total Body Clearance (CL/F) | Day 1 predose up to Day 7 postdose
Apparent Volume of Distribution During the Terminal Phase (Vz/F) | Day 1 predose up to Day 7 postdose
Area Under the Concentration-time Curve from the Time of Dosing Until the Last Measurable Concentration (AUClast) | Day 1 predose up to Day 7 postdose

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From the first dose of study drug up to 7 days postdose
  Safety is monitored by collecting AEs, which includes abnormal laboratory tests, vital signs or ECG data that are defined as an AE if the abnormality induces clinical signs or symptoms, requires active intervention, interruption or discontinuation of study medication or is clinically significant in the investigator's opinion. A treatment-emergent adverse event (TEAE) is defined as an AE that occurs or worsens after study drug administration. A serious AE (SAE) is any untoward medical occurrence that, at any dose: Results in death, is life-threatening, results in persistent or significant disability/incapacity, results in congenital anomaly, or birth defect, requires inpatient hospitalization or leads to prolongation of hospitalization or other medically important events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (7):
- Site: 3201, Ghent, Belgium
- Québec, Quebec, Canada
- Site: 4501, Århus N, Denmark
- Site: 3102, Utrecht, Netherlands
- Site: 4801, Warsaw, Poland
- Site: 90, Ankara, Turkey (Türkiye)
- Site: 44, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=245